CLINICAL TRIAL: NCT00465803
Title: Compliance Study Comparing DuoTrav to TRAVATAN Plus Timolol Using the Dosing Aid
Brief Title: A Phase IIIb Study of DuoTrav to Treat Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-06-21
Record Dates: First submitted 2007-04-23; First posted 2007-04-25 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2012-05

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
Keywords: Open-angle glaucoma or ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost; Timolol; Ophthalmic Solutions; Duotrav

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DuoTrav (Other): One drop in the study eye(s) once daily at either 8 AM or 8 PM for twelve months, as recorded by dosing aid
  Interventions: Drug: Travoprost 0.004%/timolol 0.5% ophthalmic solution
- Travatan/Timolol (Other): One drop Timolol in the study eye(s) once daily at 8 AM; one drop of Travatan in the study eye(s) once daily at 8 PM. Both products dosed for twelve months, as recorded by separate dosing aid for each product.
  Interventions: Drug: Travoprost ophthalmic solution, 0.004%; Drug: Timolol maleate ophthalmic solution, 0.5%

INTERVENTIONS:
Drug: Travoprost 0.004%/timolol 0.5% ophthalmic solution — One drop in the study eye(s) once daily at either 8 AM or 8 PM for twelve months using the Dosing Aid
  Other Names: DuoTrav
  Arms: DuoTrav
Drug: Travoprost ophthalmic solution, 0.004% — One drop in the study eye(s) once daily at 8 PM for twelve months using the Dosing Aid
  Other Names: TRAVATAN
  Arms: Travatan/Timolol
Drug: Timolol maleate ophthalmic solution, 0.5% — One drop in the study eye(s) once daily at 8 AM or twelve months using the Dosing Aid
  Arms: Travatan/Timolol

SUMMARY:
The purpose of this study is to assess patient compliance with DuoTrav versus concomitant administration of Timolol 0.5% plus TRAVATAN in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with open-angle glaucoma or ocular hypertension;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Visual acuity worse than 0.60;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2007-03; Primary Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Patient compliance | 12 months
  Patient compliance will be measured with a dosing aid that records time and date of study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Landry, Study Director — Alcon Research
Locations (1):
- Seattle, Seattle, Washington, United States